CLINICAL TRIAL: NCT04743440
Title: Bronchoscopic Endotracheal Intubation Through a Supraglottic Airway Device - an Evaluation of Physician Performance
Brief Title: Bronchoscopic Endotracheal Intubation Through a SAD - Physician Performance
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bronchoscope-sad-performance
Record Dates: First submitted 2021-01-26; First posted 2021-02-08 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2021-01

CONDITIONS: Airway Morbidity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Physicians: We will include specialists in anaesthesiology who work at the Anaesthesiology Department, Hillerød hospital, during the trial period. It is an inclusion criterion that they take part in the Anaesthesiology Department's specialist in-house on-call rotation (i.e., attending physician). Each of the included physician participants will be responsible for conducting the airway management in four patient participants; two who have been randomised to the i-gelTM LMA, and two to the Ambu® AuraGainTM LMA, respectively.
  Interventions: Device: Bronchoscopic endotracheal intubation through a supraglottic airway device

INTERVENTIONS:
Device: Bronchoscopic endotracheal intubation through a supraglottic airway device — Prior to trial commencement, participants will be asked to watch a video demonstrating preparation and conduction of the procedure (bronchoscopic endotracheal intubation through a supraglottic airway device) in a patient not involved in the project. Afterwards they will submit an online test, examining knowledge of the procedure relating to the procedure checklist. After participants have watched the demonstration video and submitted the online test, trial investigator will demonstrate the procedure in the manikin; subsequently, they have the opportunity to train the procedure in the manikin with both Igel and Auragain - training estimated to take less than 30 minutes. Afterwards, they will have the opportunity to train the procedure on manikins, on their own discretion, as per usual standards for maintaining airway competence at the Anaesthesiology Department.

SUMMARY:
Prospective observational study with the primary objective is to assess technical competence in anaesthesiology specialists who perform bronchoscopic endotracheal intubation through a supraglottic airway device (SAD), by using a global rating assessment scale (GRS) and a procedure checklist. We will use an Objective Structured Assessment of Technical Skills (OSATS)-inspired GRS that previously have been validated for fiberoptic intubation and a novel clinical checklist developed for the procedure. Secondarily, we will examine potential predictor variables.

DETAILED DESCRIPTION:
This study is a preplanned prospective observational substudy of a randomised controlled trial (RCT) with the primary aim to compare time to intubation when using two different supraglottic airway devices (SAD) as conduit for bronchoscopic intubation: the Ambu® AuraGain LMA as compared to the i-gel LMA (reference: I-gel vs AuraGain for Bronchoscopic Intubation Through SGA (ClinicalTrials.gov Identifier: NCT04680169)).

We will include all physicians who provide the airway management in the RCT.

The primary objective is to assess technical competence/performance by using a global rating assessment scale (GRS) and a procedure checklist. We will use an Objective Structured Assessment of Technical Skills (OSATS)-inspired GRS that previously have been validated for fiberoptic intubation and a novel clinical checklist developed for the procedure. Secondarily, we will examine potential predictor variables in multivariate analyses

Airway management will be video recorded. Two anaesthesiologists specialists (assessors), not otherwise involved in the trial and not employed at the hospital, will watch the video recordings of each case of airway management, i.e., the complete airway management provided by a responsible physician participant for each of the included patient participants.

For each case of airway management, they will access the physician's technical performance during the attempt to perform bronchoscopic endotracheal intubation through a SAD.

Assessors will complete a checklist during the procedure. Each item is dichotomously evaluated: done correctly (score=1)/done incorrectly or not performed (score=0). The checklist score represents the sum score for the 30 items (potential sum score range 0-30).

Assessors will evaluate the physician's technical performance using a validated GRS, scored from 8 to 40, for each case of airway management. The GRS is based on 8 items. Each item is scored from one (poor) to five (superior). A score of three is considered 'competent' for each item. The GRS score represent the sum score for all items.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthetist specialists performing bronchoskopic tracheal intubation through a supraglottic airway device
* The supraglottic airway device is either i-gelTM or a Ambu® AuraGainTM (4 in total, 2 of each i random order).

Exclusion Criteria:

* Refuse to participate
* Any other involvement in the research project

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anaesthetist specialists.It is an inclusion criterion that they take part in the anaesthesiology department's specialist in-house on-call rotation (i.e., attending physician).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Physician performance | 6 months
  Overall median physician performance score using an Objective Structured Assessment of Technical Skills (OSATS)-inspired validated global rating scale (GRS)

SECONDARY OUTCOMES:
Checklist score | 6 months
  Median checklist scores using a novel check list developed for the procedure
Pass rate | 6 months
  Overall pass rate (every item in the GRS evaluation has been scored to 3 or more)
Self-reported confidence | 6 months
  Median self-reported confidence score for the procedure during the trial (numeric rating scale (NRS) score 0-10)
GRS score progression | 6 months
  Difference in GRS scores between the first and the last patient participant (expectedly the fourth patient) in whom the physician conduct airway management.
interrater-agreement for GRS evaluation | 6 months
  interrater-agreement between assessors for the GRS evaluation

OTHER OUTCOMES:
Time to intubation | 6 months
  Time to intubation
Predictors for GRS scores | 6 months
  We will investigate the influence of the following potential predictor variables:
  Physician characteristics:
  1. Self reported experience prior to trial commencement (years since anaesthesiology specialist certification)
  2. Self-reported number of key difficult airway procedures/year in patients prior to trial commencement.
  3. Self-reported confidence for conducting the procedure, prior to trial commencement (NRS score 0-10),
  4. Number of patient participant (1-4),
  5. Type of SAD (Ambu® AuraGainTM SAD or i-gelTM SAD);
     Patient characteristics:
  6. sex,
  7. age,
  8. SARI-score
Predictors for time to intubation | 6 months
  We will investigate the influence of the following potential predictor variables:
  Physician characteristics:
  1. Self reported experience prior to trial commencement (years since anaesthesiology specialist certification)
  2. Self-reported number of key difficult airway procedures/year in patients prior to trial commencement.
  3. Self-reported confidence for conducting the procedure, prior to trial commencement (NRS score 0-10),
  4. Number of patient participant (1-4),
  5. Type of SAD (Ambu® AuraGainTM SAD or i-gelTM SAD);
     Patient characteristics:
  6. sex,
  7. age,
  8. SARI-score

CONTACTS AND LOCATIONS:
Locations (1):
- Nordsjaellands hospital Hilleroed, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No